CLINICAL TRIAL: NCT06659289
Title: Efficacy and Safety of Lipopolysaccharide Adsorption (Efferon LPS) During Cardiac Surgery Using Cardiopulmonary Bypass to Reduce the Incidence of Multiple Organ Dysfunction Syndrome in the Postoperative Period
Brief Title: Hemoperfusion Efferon LPS During Cardiac Surgery Using Cardiopulmonary Bypass
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to futility. Post-enrollment analysis of baseline disease severity indicated that the enrolled population would not allow for a meaningful assessment of the treatment effect on the primary endpoint.
Sponsor: Efferon JSC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: efferon-lps-2024-03
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Cardiac Disease; Multiple Organ Dysfunction Syndrome
Keywords: Hemoperfusion; Extracorporeal therapy; Lipopolysaccharide adsorption
MeSH Terms: conditions — Heart Diseases; Multiple Organ Failure

STUDY DESIGN:
Intervention Model Description: The study will use a 1:1 stratified randomisation. The stratification will be based on the patient's stage of CKD at the time of enrolment (strata - stages 0-2, 3-4).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline therapy (No Intervention): Patients will be treated according to the standard protocol for cardiac surgery with cardiopulmonary bypass without hemoperfusion.
- Basic therapy + Efferon LPS (Experimental): Patients will be treated according to the standard protocol for cardiac surgery with cardiopulmonary bypass and will receive hemoperfusion with Efferon LPS.
  Interventions: Device: Efferon LPS

INTERVENTIONS:
Device: Efferon LPS — Efferon LPS, a medical device, which is a single-use cartridge filled with a polymeric adsorbent that selectively adsorbs endotoxin via surface-immobilized ligand and excessive cytokines via its intrinsic porosity.
  The hemoperfusion procedure is performed at the time of cardiopulmonary bypass during cardiac surgery. The therapy (Efferon LPS hemoperfusion) is performed once. The duration of the procedure is limited by the time ofcardiopulmonary bypass.
  Arms: Basic therapy + Efferon LPS

SUMMARY:
More than 1 million people undergo cardiac surgery each year worldwide. Cardiac surgeries still in most cases require cardiopulmonary bypass, use of myocardial protection against aortic clamping and creation of cardioplegic arrest of the heart by injecting cardioplegic solutions into the coronary bed. All of the above is a source of myocardial ischemia-reperfusion injury, which remains the leading cause of acute heart failure in the period after the return of spontaneous circulation and, as a consequence, the development of post-perfusion multiple organ dysfunction syndrome and, in particular, acute kidney injury (AKI). Acute kidney injury typically develops in 7% of all hospitalised patients, 30% of intensive care unit patients and 30% of cardiac surgery patients. Endotoxemia is a major cause of AKI. Septic AKI (compared to non-septic AKI) is associated with a worse prognosis, longer hospital stay and poorer survival.

The use of the Efferon LPS hemoperfusion device, which has proven efficacy in removing not only endotoxin but also cytokines, may be promising in preventing the development of multiple organ dysfunction syndrome and in particular AKI in patients after cardiac surgery with cardiopulmonary bypass.

DETAILED DESCRIPTION:
Every year, more than 1 million people around the world undergo heart surgery. Cardiac surgery still requires cardiopulmonary bypass in the majority of cases for a number of reasons. The use of cardiopulmonary bypass in cardiothoracic surgery is a well-known and potent inducer of immune responses due to the contact of whole blood with air and extracorporeal circuit surfaces, ischemia-reperfusion injury, hemolysis and release of free hemoglobin, the effects of surgical trauma itself, and other factors.The activation of immune cells leads to the release of cytokines and inflammatory mediators such as IL-6, IL-8, activated complement and others.

One of the most common post-operative complications associated with the administration of cardiopulmonary bypass during surgery is acute kidney injury (AKI). AKI develops in 30% of patients undergoing cardiac surgery and is associated with high mortality, longer hospital stay, dialysis dependency, high risk of infectious complications and ultimately poor quality of life. Endotoxemia is a major cause of AKI. Septic AKI (compared to non-septic AKI) is associated with a worse prognosis, longer hospital stay and poorer survival.

Currently, hemosorbents based on highly cross-linked styrene/divinylbenzene copolymers can remove endo- and exotoxins in sepsis and acute and chronic renal and hepatic failure, remove intoxication by pharmacological drugs, narcotics and poisons, and remove cytokines produced in excess in systemic inflammatory syndromes of various aetiologies, including systemic inflammatory response syndrome after open-heart surgery with cardiopulmonary bypass.

Hemoperfusion is a method of extracorporeal removal of toxic substances from the blood by adsorption to a porous material. Hemoperfusion can be a good complement or substitute to the classical methods of hemofiltration and hemodialysis when diffusion or convection of toxic substances through the membrane is not efficient enough.

Based on previous studies, the use of the Efferon LPS hemoperfusion device, which has proven efficacy in removing not only endotoxin but also cytokines, may be promising in preventing the development of multiple organ dysfunction syndrome and in particular AKI in patients after cardiac surgery with cardiopulmonary bypass.

ELIGIBILITY:
Inclusion Criteria:

* Planned cardiac surgery (aortocoronary bypass, heart valve replacement, etc.) requiring the use of cardiopulmonary bypass

Exclusion Criteria:

* Emergency nature of cardiac surgery
* Cases in which a surgical procedure is required in addition to an aortocoronary artery bypass graft operation
* History of aortocoronary bypass surgery
* History of hemato-oncology
* Receiving immunosuppressive therapy for cancer and autoimmune diseases
* Sepsis, acute heart failure, acute respiratory failure, acute kidney injury at the time of enrolment
* Chronic kidney disease, stage 5D (requiring continuous hemodialysis)
* Treatment with renal replacement therapy in the past 90 days
* Presence of cirrhosis (>5 Child-Pugh score)
* Acute pulmonary embolism
* Acute myocardial infarction within 3 weeks before elective surgery
* Left ventricular ejection fraction (LVEF) less than 40% according to echocardiography
* Acute cerebrovascular accident within 3 weeks before elective surgery
* Pregnancy
* Any other clinical condition of the patient that, in the opinion of the investigator, precludes inclusion in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-04-22 (Actual); Study Completion 2025-05-06 (Actual)

PRIMARY OUTCOMES:
Effect of the hemoperfusion with Efferon LPS device during cardiopulmonary bypass on measures of organ dysfunction | 0-72 hours
  Measured every 24 hours ± 1 hour from the end of cardiopulmonary bypass to 72 hours. The SOFA (Sequential Organ Failure Assessment) index is equal to the sum of six indicators. The higher the score, the greater the insufficiency of the system being assessed. The higher the overall index, the greater the degree of multiorgan dysfunction. Violation of the function of each organ (system) is assessed separately in dynamics against the background of intensive therapy. With a score of no more than 12, multiple organ dysfunctions are assumed, 13-17 points indicate the transition of dysfunction to insufficiency, a score of about 24 indicates a high probability of death. The lower the SOFA index, the less pronounced organ failure and the better the patient's survival prognosis.

SECONDARY OUTCOMES:
Incidence of post-operative acute kidney injury | 0-72 hours
  Incidence of post-operative acute kidney injury is verified by Acute Kidney Injury Network (AKIN) criteria
Renal function | 0-72 hours
  Time (number of hours) to return to normal glomerular filtration rate (GFR)
Duration of renal replacement therapy | 1-28 days
  Duration (hours) of renal replacement therapy in patients with advanced acute kidney injury. The criteria for the end of replacement therapy is the restoration of spontaneous diuresis of more than 50 mL/hour without stimulation of diuresis with drugs or more than 2000 mL/day with stimulation.
Mean arterial pressure | 0-72 hours
  Mean arterial pressure mmHg (measured every 24 hours ±1 hour)
Duration of vasopressor support | 0-72 hours
  Time (hours) to end of vasopressor support
Pulmonary oxygen metabolic function index | 0-72 hours
  Measuring PaO2 / FiO2 index every 24 hours
Incidence of postperfusion heart failure | 0-72 hours
  Incidence of postperfusion heart failure
Duration of the need for pharmacological and/or mechanical inotropic myocardial support | 0-72 hours
  Duration (number of hours) of the need for pharmacological and/or mechanical inotropic myocardial support from the beginning of the operation to 72 hours.
Duration of ventilation | 1-14 days
  The time (hours) from the start of the operation until you are weaned off the ventilator within 14 days, or are discharged from hospital or transferred from intensive care (if earlier than day 14).
ICU length of stay | 1-14 days
  Time (days) from the end of cardiopulmonary bypass to transfer from the ICU within 14 days or hospital discharge (if earlier than day 14)
28-day mortality | Time from randomisation to 28 days from the moment of randomisation
  The number of trial participants who died in intensive care or in hospital within 28 days of randomisation
Incidence of septic complications | 1-14 days
  The number of patients who were diagnosed with sepsis after the end of cardiopulmonary bypass in the post-operative period according to the Sepsis-3 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Yuri Polushin, PhD,MD, Principal Investigator — Pavlov First Saint Petersburg State Medical University
Locations (1):
- Pavlov First Saint Petersburg State Medical University, Saint Petersburg, Russia